CLINICAL TRIAL: NCT06317363
Title: Effects of Acapella VS Chest Physiotherapy on Dyspnea, Pulmonary Functions and Air Way Clearance in Post-Operative CABG Patients
Brief Title: Effects of Acapella VS CHEST Physiotherapy in Post-Operative CABG Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0353
Record Dates: First submitted 2024-03-04; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: CABG
Keywords: Cardiac surgery; CABG; Pulmonary function; Airway clearance; Dyspnea; post-operative complications; Pneumonia; Atelectasis
MeSH Terms: conditions — Dyspnea; Pneumonia; Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group A (ACAPELLA) (Experimental): Group A (baseline treatment + acapella)
  Interventions: Other: Base Line + ACEPELLA
- Experimental Group B (MANUAL CHEST PHYSIOTHERAPY) (Experimental): Group B (baseline + manual chest physiotherapy)
  Interventions: Other: Base Line + Manual Chest Physiotherapy

INTERVENTIONS:
Other: Base Line + ACEPELLA — Group A (baseline treatment + acapella) consisting of 15 participants will receive (baseline treatment aerosol therapy, ACBT, Mobilization, breathing with arm elevation with addition to using Acapella). The primary and secondary outcome measures will be assessed at baseline post-op day 1, and after 1 week of surgery.
  Arms: Experimental Group A (ACAPELLA)
Other: Base Line + Manual Chest Physiotherapy — The group B consisting of 15 participants will receive base line treatment. aerosol therapy, ACBT, Mobilization, breathing with arm elevation with addition chest physiotherapy percussing for 20 minute. The s primary and secondary outcome measures will be assessed at baseline post-op day 1, and after 1 week of surgery.
  Arms: Experimental Group B (MANUAL CHEST PHYSIOTHERAPY)

SUMMARY:
Coronary artery bypass grafting (CABG) is a surgical procedure that is performed to improve blood flow to the heart by bypassing blocked or narrowed arteries. CABG is a major surgery that is associated with significant postoperative complications, including pulmonary complications such as atelectasis and pneumonia. Chest physiotherapy is commonly use to prevent and treat these complications, but its effectiveness in post-operative CABG patients is not well established.

The purpose of this study is to evaluate the effects of Acapella device vs chest physiotherapy on pulmonary function, airway clearance and dyspnea in post-operative CABG patients. The group A will receive (baseline treatment aerosol therapy, ACBT, Mobilization, breathing with arm elevation with addition to using Acapella), while the group B will receive base line treatment. aerosol therapy, ACBT, Mobilization, breathing with arm elevation with addition chest physiotherapy percussing for 20 minute The primary outcome measures of the study will be pulmonary function tests, including forced vital capacity (FVC), forced expiratory volume in one second (FEV1), and FEV1/FVC, and Modified Borg dyspnea scale . The secondary outcome measures will be the amount of sputum cleared. The study will be conducted over a period of 6 months after approval of synopsis.

The study will be conducted in a tertiary care hospital in Lahore, Pakistan. Patients who have undergone CABG surgery will be screen for eligibility and those who meet the inclusion criteria will be enroll in the study. Patients who have a history of chronic lung disease, smoking, intubated patient or other respiratory conditions will be exclude from the study

ELIGIBILITY:
Inclusion Criteria:

* both gender
* Patients aged between 55-70 years
* Vitally Stable
* extubated post-CABG day 01 patients
* Patient undergone for the 1st time CABG

Exclusion Criteria:

* With a history of chronic obstructive pulmonary disease or asthma patient
* Intubated patient
* Surgical complication after CABG
* With a history of smoking
* Patients who have undergone thoracic surgery in the past
* Patients with a history of neuromuscular disorders
* Patients with a history of heart failure
* Vitally unstable or on ventilator post CABG patients

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Modified Borg Dyspnea Scale | 1 week
  It is a subjective tool to assess degree of dyspnea in patients. The comprise of 10 grades starting from zero to 10. Zero refers to 'No difficulty in breathing at all 'and 10 refers to 'maximal difficulty ' Readings will be taken at 1st post op day and after post op week 1
FEV1 | 1 week
  digital spirometer device will be used to take readings of lung volumes in (ml). These measurements are part of a pulmonary function test, which helps diagnose and monitor respiratory conditions such as asthma, chronic obstructive pulmonary disease (COPD), and cystic fibrosis. Readings will be taken at 1st post op day and after 1st post op week
FVC | 1 week
  digital spirometer device will be used to take readings of lung capacities in (ml). These measurements are part of a pulmonary function test, which helps diagnose and monitor respiratory conditions such as asthma, chronic obstructive pulmonary disease (COPD), and cystic fibrosis. Readings will be taken at 1st post op day and after 1st post op week
FEV1/FVC | 1 week
  digital spirometer device will be used to take readings of FEV1/FVC. Readings will be taken at 1st post op day and after 1st post op week
sputum volume | 1 Weeks
  A sputum collection jar will be used to record the amount of sputum produced by a patient over a specific period of time in (ml). Sputum is a mixture of saliva and mucus that is expectorated from the lungs. By tracking the amount and consistency of sputum, healthcare professionals can monitor the progression of respiratory conditions and assess the effectiveness of treatment.
  The readings of these outcome measure will be taken two times. 1st post op day and after 1st week

SECONDARY OUTCOMES:
body temperature(degree centigrade) | 1 week
  Pre-post readings of vitals will be taken from monitor attached to the patient
pulse rate (beats/minute) | 1 week
  Pre-post readings of vitals will be taken from monitor attached to the patient
respiratory rate( breaths/minute) | 1 week
  Pre-post readings of vitals will be taken from monitor attached to the patient
blood pressure (mmHg) | 1 week
  Pre-post readings of vitals will be taken from monitor attached to the patient
SpO2 (%) | 1 week
  pre-post readings will be taken of oxygenic indicators through ABGs
SaO2 (%) | 1 week
  pre-post readings will be taken of oxygenic indicators through ABGs
PaO2 (%) | 1 week
  pre-post readings will be taken of oxygenic indicators through ABGs
PaCO2 (%) | 1 week
  pre-post readings will be taken of oxygenic indicators through ABGs

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Muriam Ghani, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farina P, Gaudino MFL, Taggart DP. The Eternal Debate With a Consistent Answer: CABG vs PCI. Semin Thorac Cardiovasc Surg. 2020 Spring;32(1):14-20. doi: 10.1053/j.semtcvs.2019.08.009. Epub 2019 Aug 20. PMID 31442489
- [Background] Jannati M, Navaei MR, Ronizi LG. A comparative review of the outcomes of using arterial versus venous conduits in coronary artery bypass graft (CABG). J Family Med Prim Care. 2019 Sep 30;8(9):2768-2773. doi: 10.4103/jfmpc.jfmpc_367_19. eCollection 2019 Sep. PMID 31681641
- [Background] Shawon MSR, Odutola M, Falster MO, Jorm LR. Patient and hospital factors associated with 30-day readmissions after coronary artery bypass graft (CABG) surgery: a systematic review and meta-analysis. J Cardiothorac Surg. 2021 Jun 10;16(1):172. doi: 10.1186/s13019-021-01556-1. PMID 34112216
- [Background] Yamamoto K, Natsuaki M, Morimoto T, Shiomi H, Matsumura-Nakano Y, Nakatsuma K, Watanabe H, Yamamoto E, Kato E, Fuki M, Yamaji K, Nishikawa R, Nagao K, Takeji Y, Watanabe H, Tazaki J, Watanabe S, Saito N, Yamazaki K, Soga Y, Komiya T, Ando K, Minatoya K, Furukawa Y, Nakagawa Y, Kadota K, Kimura T; CREDO-Kyoto PCI/CABG Registry Cohort-3 investigators. Periprocedural Stroke After Coronary Revascularization (from the CREDO-Kyoto PCI/CABG Registry Cohort-3). Am J Cardiol. 2021 Mar 1;142:35-43. doi: 10.1016/j.amjcard.2020.11.031. Epub 2020 Dec 3. PMID 33279479
- [Background] Rupprecht L, Schmid C, Debl K, Lunz D, Florchinger B, Keyser A. Impact of coronary angiography early after CABG for suspected postoperative myocardial ischemia. J Cardiothorac Surg. 2019 Mar 12;14(1):54. doi: 10.1186/s13019-019-0876-0. PMID 30871615
- [Background] Moradian ST, Heydari AA, Mahmoudi H. What is the Role of Preoperative Breathing Exercises in Reducing Postoperative Atelectasis after CABG? Rev Recent Clin Trials. 2019;14(4):275-279. doi: 10.2174/1574887114666190710165951. PMID 31291879
- [Background] Chen X, Li C, Zeng L, Rong T, Lin P, Wang Q, Guo Z, Long H, Zhong J. Comparative efficacy of different combinations of acapella, active cycle of breathing technique, and external diaphragmatic pacing in perioperative patients with lung cancer: a randomised controlled trial. BMC Cancer. 2023 Mar 28;23(1):282. doi: 10.1186/s12885-023-10750-4. PMID 36978035